CLINICAL TRIAL: NCT05630859
Title: A Phase 1/2, Observer-blind, Randomized, Placebo-controlled Multi-country Study to Assess Safety and Efficacy of GSK Neisseria Gonorrhoeae GMMA (NgG) Investigational Vaccine When Administered to Healthy Adults 18 to 50 Years of Age
Brief Title: Safety and Efficacy of GSK Neisseria Gonorrhoeae GMMA (NgG) Investigational Vaccine When Administered to Healthy Adults 18 to 50 Years of Age.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 216156; 2022-500883-37-00 (Other: EU CT number)
Record Dates: First submitted 2022-11-25; First posted 2022-11-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Sexually Transmitted Diseases
Keywords: Neisseria gonorrhoeae; Safety; Efficacy; Sexually transmitted infection; Healthy adults 18 to 50 years of age
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Phase 1:1a Low dose Group (Experimental): Participants randomized to the 1a Low dose Group receive 2 doses of NgG low dose investigational vaccine.
  Interventions: Biological: NgG low dose investigational vaccine
- Phase 1:1b Placebo Group (Placebo Comparator): Participants randomized to the 1b Placebo Group receive 2 doses of placebo.
  Interventions: Biological: Placebo
- Phase 1: 2a Medium dose Group (Experimental): Participants randomized to the 2a Medium dose Group receive 2 doses of NgG medium dose investigational vaccine.
  Interventions: Biological: NgG medium dose investigational vaccine
- Phase 1: 2b Placebo Group (Placebo Comparator): Participants randomized to the 2b Placebo Group receive 2 doses of placebo.
  Interventions: Biological: Placebo
- Phase 1: 3a High dose Group (Experimental): Participants randomized to the 3a High dose Group receive 2 doses of NgG high dose investigational vaccine.
  Interventions: Biological: NgG high dose investigational vaccine
- Phase 1: 3b Placebo Group (Placebo Comparator): Participants randomized to the 3b Placebo Group receive 2 doses of placebo.
  Interventions: Biological: Placebo
- Phase 2: 4a HTD Group (Experimental): Participants randomized to the 4a highest tolerated dose (HTD) Group receive 2 doses of NgG highest tolerated dose selected from Phase 1.
  Interventions: Biological: NgG HTD investigational vaccine
- Phase 2: 4b dose below HTD Group (Experimental): Participants randomized to the 4b dose below HTD Group receive 2 doses of NgG dose below the highest tolerated dose selected from Phase 1.
  Interventions: Biological: NgG below HTD investigational vaccine
- Phase 2: 4c Placebo Group (Placebo Comparator): Participants randomized to the 4c Placebo Group receive 2 doses of placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NgG low dose investigational vaccine — Two doses of NgG low dose investigational vaccine, administered intramuscularly.
  Arms: Phase 1:1a Low dose Group
Biological: NgG medium dose investigational vaccine — Two doses of NgG medium dose investigational vaccine, administered intramuscularly.
  Arms: Phase 1: 2a Medium dose Group
Biological: NgG high dose investigational vaccine — Two doses of NgG high dose investigational vaccine, administered intramuscularly.
  Arms: Phase 1: 3a High dose Group
Biological: Placebo — Two doses of placebo, administered intramuscularly.
  Other Names: Sodium chloride (NaCl)
  Arms: Phase 1: 2b Placebo Group; Phase 1: 3b Placebo Group; Phase 1:1b Placebo Group; Phase 2: 4c Placebo Group
Biological: NgG HTD investigational vaccine — Two doses of NgG HTD investigational vaccine, administered intramuscularly.
  Arms: Phase 2: 4a HTD Group
Biological: NgG below HTD investigational vaccine — Two doses of NgG below HTD investigational vaccine, administered intramuscularly.
  Arms: Phase 2: 4b dose below HTD Group

SUMMARY:
The aim of this first time in human proof of concept (FTiH-PoC) study is to evaluate safety and reactogenicity, to demonstrate efficacy and to explore immunogenicity of GlaxoSmithKline's (GSK) Neisseria gonorrhoeae generalized modules for membrane antigens (GMMA) (NgG) investigational vaccine compared to placebo (saline).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the dose-escalation safety lead-in part

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history, clinical examination, and laboratory assessment.
* A participant between and including 18 and 50 years of age at the time of informed consent.
* Female participants of non-childbearing potential may be enrolled in the study.
* Female participants of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration series.

Inclusion criteria for the efficacy PoC part

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by:

  * For the 2 intensive safety monitoring subsets (i.e., first 30 HIV negative subjects per group followed by first 8 HIV positive subjects per group): medical history, clinical examination, and laboratory assessment.
  * For all the remaining participants: medical history, clinical examination.
* At risk for gonococcus infections based on sexual behavioral characteristics: this may include men having sex with men, pre-exposure prophylaxis for HIV users, individuals who engage in transactional sex participants with current or past STI diagnosis, participants at time of STI screening or seeking other STI services.
* A participant between and including 18 and 50 years of age at the time of informed consent. Transgender men and women, and other gender non-conforming people who identify themselves as neither men nor women may be enrolled into the study, based on their risk factors. For the purpose of this study, they will be followed up according to their biological sex (sex at birth), sexual orientation, and genital/sexual anatomy
* Participants of non-childbearing potential may be enrolled in the study. This includes transmen that have not undergone gender affirming surgery of their genitals.
* Participants of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration series.

Exclusion criteria:

1. Medical conditions Dose-escalation safety lead-in part

   * Any clinically significant biochemical laboratory abnormality.
   * Any other clinical condition as determined by the investigator, that may increase participant's risk due to study participation.
   * History of any reaction/hypersensitivity likely to be exacerbated by any component of the study intervention.
   * Confirmed or suspected immunosuppressive/immunodeficient condition, based on medical history and physical examination.
   * Hypersensitivity to latex.
   * Acute/chronic clinically significant pulmonary, cardiovascular, hepatic/renal functional abnormality, as determined by physical examination/laboratory tests.
   * Uncontrolled neurological disorders or seizures.
   * History of invasive meningococcal disease. Efficacy PoC part: HIV negative intensive safety monitoring, HIV negative full enrollment and for all remaining participants
   * Persons under guardianship or trusteeship.
   * Persons deprived of liberty.
   * Gonococcal infection identified within 14 days prior to randomization.
   * Any other clinical condition as determined by the investigator, that may increase participant's risk due to study participation.
   * History of severe allergic reactions and/anaphylaxis, or any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
   * Bleeding diathesis / any other condition that would contraindicate intramuscular administration.
   * Confirmed or suspected immunosuppressive/immunodeficient condition, based on medical history and physical examination.
   * Known seropositivity for HIV infection, regardless of viremia and CD4 cell count
   * Hypersensitivity to latex.
   * Acute/chronic clinically significant pulmonary, cardiovascular, hepatic/renal functional abnormality, as determined by physical examination/laboratory tests.
   * Recurrent history/uncontrolled neurological disorders or seizures.
   * History of invasive meningococcal disease.

   The exclusion criteria depicted above, and the following exclusions criterion applies only for the HIV positive participants (intensive safety monitoring subset and full enrollment of HIV positive participants):

   Seropositivity for HIV infection if:
   * CD4 cell count < 350 cells/mm3 in the last 6 months
   * viral load > 50cp/ml in the last 6 months
   * participant is not on antiretroviral therapy (ART) for > 3 months or has switched from a different ART in the last 3 months.

   For both Intensive safety monitoring subset (first 30 HIV negative subjects per group and first 8 HIV positive subjects per group) these criteria apply:

   Any clinically significant hematological/biochemical laboratory abnormality.
2. Prior/Concomitant therapy Applicable for both the dose-escalation safety lead-in part and the PoC part

   * Use of any investigational/non-registered product other than the study intervention(s) within 30 days before the first dose/planned use during the study period.
   * Previous and planned vaccination with an OMV based Neisseria meningitidis group B vaccine (e.g., Bexsero, MeNZB vaccine or MenBvac at any time prior to first dose and during the entire study period.
   * Planned administration/administration of a vaccine not specified in study protocol within 15 days before the first dose and ending 15 days after the last dose of vaccine administration.
   * Administration of long-acting immune-modifying drugs during the period starting 6 months prior to the first dose of study intervention/planned administration at any time during the study period.
   * Administration of immunoglobulins /any blood products/plasma derivatives during the period starting 3 months before the administration of the first dose of study intervention/planned administration during the study period.
   * Chronic administration (more than 14 days in total) of immunosuppressants/other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose(s). For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants/ ≥0.5 mg/kg/day. Inhaled and topical steroids are allowed.

   The following criterion applies only for the PoC part:

   •Chronic/long-term use of systemic antibiotics with an activity against Neisseria gonorrhoeae.
3. Prior/Concurrent clinical study experience applicable for both dose-escalation safety lead-in part and the PoC part Concurrently participating in another clinical study, at any time during the study period, in which the participant has been/will be exposed to an investigational/a non-investigational intervention.
4. Other exclusions applicable for both dose-escalation safety leading part and the PoC part

   * Pregnant/lactating female.
   * Female planning to become pregnant/to discontinue contraceptive precautions before 1 month after completion of the study intervention administration series.
   * Any study personnel/their immediate dependents, family/household members.
   * Lifestyle consideration that may interfere with the conduct of the study/pose additional risks to the rights and wellbeing of participants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1004 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting solicited administration site events in study Phase 1 (Dose-escalation safety lead-in) | During the 7 days follow-up period after the first dose
  The solicited administration site events after vaccination include pain, redness, and swelling.
Percentage of participants reporting solicited administration site events in study Phase 1 (Dose-escalation safety lead-in) | During the 7 days follow-up period after the second dose
  The solicited administration site events after vaccination include pain, redness, and swelling.
Percentage of participants reporting each solicited systemic event in study Phase 1 (Dose-escalation safety lead-in) | During the 7 days follow-up period after the first dose
  The solicited systemic events after vaccination include fever, headache, myalgia, arthralgia, fatigue. Fever is defined as temperature ≥38.0°C/100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
Percentage of participants reporting each solicited systemic event in study Phase 1 (Dose-escalation safety lead-in) | During the 7 days follow-up period after the second dose
  The solicited systemic events after vaccination include fever, headache, myalgia, arthralgia, fatigue. Fever is defined as temperature ≥ 38.0°C/100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
Percentage of participants reporting unsolicited adverse events (AEs) in study Phase 1 (Dose-escalation safety lead-in) | During the 30 days follow-up period after the first dose
  Any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of participants reporting unsolicited AEs in study Phase 1 (Dose-escalation safety lead-in) | During the 30 days follow-up period after the second dose
  Any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of participants reporting serious adverse events (SAEs) in study Phase 1 (Dose-escalation safety lead-in) | From Day 1 after the first dose up to study Phase I end (Day 241)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in an abnormal pregnancy outcome.
Percentage of participants reporting AEs leading to withdrawal in study Phase 1 (Dose-escalation safety lead-in) | From Day 1 after the first dose up to study Phase I end (Day 241)
  An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention.
Percentage of participants with haematological and biochemical laboratory abnormalities in study Phase 1 (Dose-escalation safety lead-in) | 7 days after the first dose
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of participants with haematological and biochemical laboratory abnormalities in study Phase 1 (Dose-escalation safety lead-in) | 7 days after the second dose
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Incidence rates of confirmed gonorrhea cases in study Phase 2 [Efficacy Proof of Concept (PoC)] | From 1 month to 13 months post-Dose 2
Percentage of participants reporting solicited administration site events in study Phase 2 (Efficacy PoC) | During the 7 days follow-up period after the first dose
  The solicited administration site events after vaccination include pain, redness, and swelling.
Percentage of participants reporting solicited administration site events in study Phase 2 (Efficacy PoC) | During the 7 days follow-up period after the second dose
  The solicited administration site events after vaccination include pain, redness, and swelling.
Percentage of participants reporting each solicited systemic event in study Phase 2 (Efficacy PoC) | During the 7 days follow-up period after the first dose
  The solicited systemic events after vaccination include fever, headache, myalgia, arthralgia, fatigue. Fever is defined as temperature ≥ 38.0°C/100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
Percentage of participants reporting each solicited systemic event in study Phase 2 (Efficacy PoC) | During the 7 days follow-up period after the second dose
  The solicited systemic events after vaccination include fever, headache, myalgia, arthralgia, fatigue. Fever is defined as temperature ≥ 38.0°C/100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
Percentage of participants reporting unsolicited AEs in study Phase 2 (Efficacy PoC) | During the 30 days follow-up period after the first dose
  Any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of participants reporting unsolicited AEs in study Phase 2 (Efficacy PoC) | During the 30 days follow-up period after the second dose
  Any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of participants reporting SAEs in study Phase 2 (Efficacy PoC) | From Day 1 after the first dose up to study end (Day 451)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in an abnormal pregnancy outcome.
Percentage of participants reporting AEs leading to withdrawal in study Phase 2 (Efficacy PoC) | From Day 1 after the first dose up to study end (Day 451)
  An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention.
Percentage of participants with haematological and biochemical laboratory abnormalities in study Phase 2 (Efficacy PoC) | 7 days after the first dose
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participants condition. The evaluation of the endpoint will be assessed in the subsets for intensive safety monitoring.
Percentage of participants with haematological and biochemical laboratory abnormalities in study Phase 2 (Efficacy PoC) | 7 days after the second dose
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.

SECONDARY OUTCOMES:
Incidence rates of confirmed gonorrhea cases with and without co-infection with a different sexually-transmitted disease causing bacterium in study Phase 2 (Efficacy PoC) | From 1 month to 13 months post-Dose 2
Incidence rates of gonorrhea in study Phase 2 (Efficacy PoC) | From 1 month to 13 months post-Dose 2
Incidence rates of other gonococcal infection with positive Ng in study Phase 2 (Efficacy PoC) | From 1 month to 13 months post-Dose 2

CONTACTS AND LOCATIONS:
Locations (21):
- United States (7):
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Austin, Texas
- GSK Investigational Site, Salvador, Brazil
- France (3):
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
- Germany (3):
  - GSK Investigational Site, Bochum
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Manila, Philippines
- South Africa (2):
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Soweto
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.